CLINICAL TRIAL: NCT00854997
Title: The Impact of Obstructive Sleep Apnea on the Outcomes in Patients of First-Time Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Peilin Lee, National Taiwan University Hospital
Other Study IDs: 200812080R
Record Dates: First submitted 2009-01-12; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Sleep Apnea, Obstructive; Acute Myocardial Infarction
Keywords: Obstructive sleep apnea; myocardial infarction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, RNA, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: AMI with OSA
- 2: AMI without OSA

SUMMARY:
Objective: Untreated OSA is associated with three fold risk of fetal and non-fetal cardiovascular events than control subjects in the long-term follow up. However, the prevalence rate and impact of OSA in patients with acute myocardial infarction (AMI) was not clear so far. The conflicts of studies come from variable period of AMI, heart function at enrollment, techniques used to diagnose OSA, time to revascularization, and target endpoint. Therefore, this project aimed to study the patients of first-time, Killip I-II, and post primary percutaneous coronary intervention (PCI) AMI in both and chronic phase to achieve four goals:

Aim 1. To determine the prevalence rate of OSA in patients with first-time AMI The acute phase of AMI was defined as within 14 days of the onset of AMI and the chronic phase was defined as > 14 days of onset. Eligible patients were screened with polysomnography within 5th to 7th days and 6th months of AMI to determine the prevalence rate of OSA in the AMI. Patients who had AHI more than 15/hr were considered as suffering from OSA.

Aim 2. To identify the clinical characteristics and risk factors in AMI patients associated with OSA Patients were followed up at clinics for five years. The baseline demographics of patients with or without OSA were compared to determine the factors associated with OSA in AMI patients.

Aim 3. To study the impact of OSA on the prognosis of AMI patients after revascularizaton The primary endpoint was mortality rate and cardiac events. The secondary endpoint was left ventricular function and variables related to cardiovascular disease (CVD) and metabolic syndrome. The impact of OSA on AMI was determined by comparing primary and secondary endpoint between AMI patients with and without OSA.

Aim 4. To identify the clinical and molecular factors attributing to AMI in OSA patients Factors attributing to AMI in OSA patients were determined by comparing the clinical data and mRNA expression of angiogenesis and other related genes in OSA patients with the acute phase of AMI and patients without major CVD.

DETAILED DESCRIPTION:
Objectives: Obstructive sleep apnea (OSA) affects 4% middle-aged men and 2% women. Symptoms of OSA include snore, unrefresh sleep, witnessed apnea, excessive daytime sleepiness and hypertension. Untreated OSA patients are associated with three fold risk of fetal and non-fetal cardiovascular events than control subjects. However, the prevalence rate and impact of OSA in patients with acute myocardial infarction (AMI) was not clear so far. The conflicts of studies come from variable period of AMI, heart function at enrollment, techniques used to diagnose OSA, time to revascularization, and target endpoint. Therefore, this project aimed to achieve the four goals: (1) To determine the prevalence rate of OSA in patients with first-time AMI (2) To identify the clinical characteristics and risk factors in AMI patients associated with OSA (3) To study the impact of OSA on the prognosis of AMI patients after revascularization (4) To identify the clinical and molecular factors attributing to AMI in OSA patients Study design: Longitudinal, observational study Participants: AMI patients who were first-time, Killip I-II, post primary percutaneous coronary intervention (PCI) were eligible for this study. Exclusion criteria included: refuse to participate, require mechanical ventilation, active neurologic event, chronic pulmonary disease, active infection, need sedatives or narcotics within 3 days of sleep study, and participate in other study at the same time.

Protocol: Eligible patients were screened with polysomnography (PSG) within 5th to 7th days after onset of AMI. Patients who had AHI more than 15/hr were considered as suffering from OSA. Patients were followed up for five years. The primary endpoint was mortality rate and cardiac events. The secondary endpoint was left ventricular function and variables related to cardiovascular disease (CVD) and metabolic syndrome. The acute phase of AMI was defined as within 14 days of the onset of AMI and the chronic phase was defined as > 14 days of onset.

Statistic: The baseline demographics of patients with or without OSA were compared to determine the factors associated with OSA in AMI patients. The impact of OSA on AMI in acute and chronic phase was determined by comparing the mortality rate, incidences of cardiac events, left ventricular function, CVD risk factors, and metabolic profiles between AMI patients with and without OSA. Factors attributing to AMI in OSA patients were determined by comparing the clinical data and mRNA expression of angiogenesis and other related genes in OSA patients with the acute phase of AMI and patients without major CVD.

Clinical implication: Because the prevalence rate of OSA in patients of first-time AMI but no significant heart failure was extremely high, early PSG screening and identifying factors associated with OSA will allow for early diagnosis and intervention. Understanding interaction between OSA and AMI will help prevent the morbidity and mortality in AMI patients. Also, it allows for prediction of cardiovascular outcomes and early management in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* first-time, Killip I-II, post primary PCI within 5th -7th day of AMI

Exclusion Criteria:

* refuse to participate, require mechanical ventilation, active neurologic event, chronic pulmonary disease, active infection, need sedatives or narcotics within 3 days of sleep study, and participate in other study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: first-time, Killip I-II, post primary PCI within 5th -7th day of AMI
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 36 months

SECONDARY OUTCOMES:
left ventricular function and variables related to cardiovascular disease (CVD) and metabolic syndrome. | 36months

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan